CLINICAL TRIAL: NCT01714336
Title: Is Tranexamic Acid Effective in Limiting Transfusion After Hip Replacement for Femoral Neck Fracture: A Randomized Controlled Trial
Brief Title: Does Tranexamic Acid Reduce the Need for Blood Transfusions in Patients Undergoing Hip Fracture Surgery?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Pagnano, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-004599
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Hip Fracture
Keywords: Arbeitsgemeinschaft für Osteosynthesefragen (AO) fracture; Orthopaedic Trauma Association (OTA) fracture
MeSH Terms: conditions — Hip Fractures; Fractures, Bone | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Normal saline will be administered intravenously in two doses of 15 mg/kg each administered over a period of ten minutes, one dose just prior to incision and the second at initiation of wound closure.
  Interventions: Drug: placebo
- tranexamic acid (Active Comparator): Tranexamic acid will be administered intravenously in two doses of 15 mg/kg each administered over a period of ten minutes, one dose just prior to incision and the second at initiation of wound closure.
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — Tranexamic acid will be administered intravenously in two doses of 15 mg/kg. Each dose will be administered over a period of ten minutes, one dose just prior to incision and the second at initiation of wound closure.
  Arms: tranexamic acid
Drug: placebo — A similar dose of 0.9% sodium chloride (NaCL) will be administered intravenously in two doses over a ten minute period, one dose at incision and the other at initiation of wound closure.
  Arms: placebo

SUMMARY:
Does tranexamic acid improve the perioperative care of those patients treated surgically for hip fracture by decreasing the proportion of patients requiring transfusion and decreasing total perioperative bleeding.

DETAILED DESCRIPTION:
Antifibrinolytic medications such as tranexamic acid, aprotinin, and aminocaproic acid have proven to be useful in decreasing blood loss and the proportion of patients who require transfusion after a number of surgical procedures. In orthopedic surgery, tranexamic acid (TXA) is the best studied of these medications and a recent Cochrane Database review determined that tranexamic acid was effective in decreasing perioperative bleeding and post-operative transfusion after elective hip replacement and knee replacement surgery. At Mayo Clinic Rochester, the routine administration of tranexamic acid has evolved over the past decade to become part of the typical protocol for more than 3,000 elective hip and knee replacement procedures each year. Recent administrative data provides fairly compelling evidence of the efficacy of tranexamic acid in decreasing transfusion at the Mayo Clinic Rochester practice with 2010 data showing 2% and 7% prevalence of transfusion in patients treated with tranexamic acid versus 18% and 33% prevalence in those knee and hip replacement patients, respectively, who were not treated with tranexamic acid. A recent analysis of the Mayo Clinic Rochester orthopedic practice showed that patients treated for hip fracture remain at substantial risk of perioperative transfusion (30% prevalence) after operative management. This raises the question as to whether tranexamic acid could improve the perioperative care of those patients treated surgically for hip fracture by decreasing the proportion of patients requiring transfusion and decreasing total perioperative bleeding.

ELIGIBILITY:
Inclusion criteria

* AO/OTA (Orthopedic Trauma Association) fracture classification 31B
* Surgically treated with either hemiarthroplasty or total hip arthroplasty
* Acute fracture treated within 72 hours of injury
* Low energy isolated injury
* Age greater than 18 years old

Exclusion Criteria

* Transfusion received during admission, prior to surgery
* Creatinine clearance less than 30 mL/min
* History of unprovoked Venous Thromboembolism (VTE) and/or recurrent VTE
* Known history of Factor V Leiden, protein C/S deficiency, prothrombin gene mutation, anti-thrombin deficiency, anti-phospholipid antibody syndrome, lupus anticoagulant
* Pregnancy or breastfeeding (pregnancy tests will be performed on all patients of child-bearing potential)
* History of cerebrovascular accident (CVA), Myocardial infarction (MI), or VTE within the previous 30 days
* Coronary stent placement within the previous 6 months
* Disseminated intravascular coagulation
* Subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pagnano, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tranexamic Acid
Started | 69 | 69
Completed | 69 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Normal saline will be administered intravenously in two doses of 15 mg/kg each administered over a period of ten minutes, one dose just prior to incision and the second at initiation of wound closure.
  placebo: A similar dose of 0.9% NaCL will be administered intravenously in two doses over a ten minute period, one dose at incision and the other at initiation of wound closure.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tranexamic Acid | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.2 (10) | 81.0 (10) | 81.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received a Hospitalization Transfusion
Description: Proportion of patients transfused at least 1 unit of packed red blood cells during hospital admission
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 18 | 12

2. Secondary Outcome: Mean Number of Units Transfused
Description: Mean number of units transfused per patient
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: units/participant transfused
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
units/participant transfused | 1.8 (0.9) | 1.2 (0.5)

3. Secondary Outcome: Calculated Blood Loss
Description: Calculated blood loss
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
cc | 1214 (540) | 902 (439)

4. Secondary Outcome: Number of Participants With Venous Thromboembolism (VTE) Diagnosis
Description: Incidence of symptomatic VTE diagnosed within 6 months of surgery
Time Frame: Within 6 months of surgery
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 2 | 3

5. Secondary Outcome: Number of Participants With Wound Complications
Description: Wound complications diagnosed within 6 months of surgery
Time Frame: Within 6 months of surgery
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 2 | 5

6. Secondary Outcome: Number of Participants With Myocardial Infarction (MI) Diagnosis
Description: MI diagnosed within 6 months of surgery
Time Frame: Within 6 months of surgery
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 3 | 2

7. Secondary Outcome: Number of Participants With Cerebrovascular Accident (CVA) Diagnosis
Description: CVA diagnosed within 6 months of surgery
Time Frame: Within 6 months of surgery
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 0 | 1

8. Secondary Outcome: Number of Participants Who Died
Description: All-cause mortality at 6 months
Time Frame: 6 months after surgery
Measure: Number; unit: participants
Arm/Group | Placebo | Tranexamic Acid
Number analyzed (Participants) | 69 | 69
participants | 11 | 10
Statistical Analysis 1: Comparison: Placebo vs Tranexamic Acid; Test type: Superiority or Other; p = 0.75, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | Placebo | Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 15/69 | 14/69
Other Adverse Events (participants affected / at risk) | 9/69 | 15/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Tranexamic Acid (N=69)
MI (Cardiac disorders) | 3 (3) | 2 (2)
CVA (Nervous system disorders) | 0 (0) | 1 (1)
Death (Surgical and medical procedures) | 6 (6) | 7 (7)
VTE (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=69) | Tranexamic Acid (N=69)
Readmission (Surgical and medical procedures) | 9 (9) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No